CLINICAL TRIAL: NCT06411756
Title: Physical Activity Intervention Co-created and Tested With African American Colorectal Cancer Survivors
Brief Title: Physical Activity Centers Empowerment
Acronym: PACE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: UNC Lineberger Comprehensive Cancer Center (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: LCCC2143AIM2; 1K23MD015719-01 (NIH)
Record Dates: First submitted 2024-05-06; First posted 2024-05-13 (Actual); Last update posted 2026-01-06 (Actual); Status verified 2026-01

CONDITIONS: Colorectal Neoplasms
Keywords: Physical activity; Colorectal Neoplasms; Health Equity; Black or African American
MeSH Terms: conditions — Colorectal Neoplasms; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Arm (Other): Subjects will receive access to the video library, a Fitbit, a daily adaptive step goal that will be sent via text message with a short positive message; and monthly Zoom meetings, led by the research team, to discuss physical activity with other study subjects.
  Interventions: Behavioral: Narrative videos; Behavioral: A Fitbit activity tracker; Other: Daily text message; Other: Monthly Zoom meeting; Other: Website access
- Control Arm (Other): Subjects will receive access to the video library after the study period (after the 9-month assessment).
  Interventions: Behavioral: A Fitbit activity tracker; Other: Printed materials; Behavioral: Printed materials

INTERVENTIONS:
Behavioral: Narrative videos — Culturally targeted narrative videos will be sent via email.
  Arms: Intervention Arm
Behavioral: A Fitbit activity tracker — A Fitbit activity tracker is a wireless wearable device that monitors physical fitness activity.
Other: Daily text message — A daily adaptive step goal that will be sent via text message with a short positive message.
  Arms: Intervention Arm
Other: Monthly Zoom meeting — Monthly Zoom meetings, led by the research team, to discuss physical activity with other study subjects.
  Arms: Intervention Arm
Other: Website access — Access to Physical Activity Centers Empowerment (PACE) website.
  Arms: Intervention Arm
Other: Printed materials — Printed materials from the American College of Sport's Medicine's "Moving through Cancer" campaign.
  Arms: Control Arm
Behavioral: Printed materials — Printed materials from the American College of Sports Medicine's "Moving through Cancer" campaign.
  Arms: Control Arm

SUMMARY:
This research study tests the feasibility of the Physical Activity Centers Empowerment (PACE) physical activity intervention for African American individuals diagnosed with colorectal cancer.

Feasibility will be measured as intervention reach, effectiveness, adoption, implementation, and maintenance. Seventy-two subjects will be recruited to conduct a pilot two-group, randomized repeated measures study.

DETAILED DESCRIPTION:
The purpose of this research is to improve the quality of life for underserved cancer survivors by increasing physical activity. A physical activity intervention will be tested for feasibility with African American cancer survivors. The project will serve as a foundation for intervening with other underserved cancer survivors.

Feasibility will be measured as intervention Reach, Effectiveness, Adoption, Implementation, and Maintenance, following the RE-AIM framework. Survey and biomarker data will be collected at baseline, 3 and 9 months later. These time points will facilitate exploration of changes pre- and post-intervention, and to determine if effects are maintained 6 months after completing the intervention. Our primary hypothesis is that the intervention will be feasible to deliver.

ELIGIBILITY:
Inclusion Criteria:

1. self-identifying as AA of Black,
2. diagnosis of CRC,
3. scheduled to receive chemotherapy,
4. age 18 years or older,
5. no contraindications to unsupervised PA as determined by the PA readiness questionnaire,
6. oncologist approval to participate, and
7. a smartphone for Fitbit syncing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2024-08-14 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Feasibility Reach- Recruitment | 18 months
  Feasibility Reach- Recruitment is measured by the number of participants screened, ineligible, eligible, enrolled and declined participation.
Feasibility Retention | 18 months
  Retention is measured by the frequency of enrolled participants continued study interventions
Average weekly steps | 3 months
  Average weekly steps and the frequency of participants achieving daily step goals. Daily steps are collected via Fitbit Inspire activity tracker. Differences in daily steps and the frequency of meeting daily step goals between the intervention and control arms.
Weekly participation in mild, moderate, and vigorous exercise | 3 months
  Weekly participation in mild, moderate, and vigorous exercise is time spent on physical activity each week is measured subjectively using the Godin Leisure-time Exercise Questionnaire (GLTEQ) and objectively by the Fitbit Inspire activity tracker. The GLTEQ asks participants to self-report how many times they do strenuous, moderate, and mild or light exercise each week and the average duration of exercise. The intervention effectiveness is operationalized by the differences in minutes of doing mild, moderate, and vigorous physical activity between the intervention and control arms.
Daily engagement in sedentary behaviors | 3 months
  Daily engagement in sedentary behaviors will be measured as time spent on sedentary behaviors per day is measured subjectively by a 10-option Likert scale called the Sedentary Behavior Questionnaire. Participants are asked to select one of the following options: none,<=15 minutes, 30 minutes,1 hour,2 hours,3 hours, 4 hours, 5 hours, and 6 hours or more" to estimate the time they spend doing each sedentary behavior on a typical week and a typical weekend day. The behaviors include watching television, playing computer or video games, sitting and listening to music on the radio, tapes, or CDs, sitting and talking on the phone, doing paperwork or computer work, sitting and reading a book or magazine, playing a musical instrument, doing artwork or crafts, and sitting and driving a car, bus or train. The total daily sedentary score ranges from 0 to 81. Daily sedentary time is also recorded objectively by the Fitbit Inspire activity tracker.
Adaption of the study | Up to 18 months
  Adaption of the study will be measured by the percentage of contacted individuals who meet study criteria to participate in the study.
Implementation of the video library | Up to 3 months
  Implementation of the video library: The percentage of participants who watched study-related video content.
Implementation of using FITBIT | Up to 3 months
  Implementation of using FITBIT: The percentage of days that participants wear the study-issued Fitbits.
The differences between intervention and control arms | 3 months to 9 months
  The Maintenance will be measured as the differences in intervention effects between intervention and control arms groups 6 months post-intervention (9 months post-baseline).

SECONDARY OUTCOMES:
Outcome expectations | Baseline, 3 months, 9 months
  Outcome expectations will be measured using the modified Multidimensional Outcome Expectations for Exercise Scale, which has an internal consistency of 0.82, 0.84, and 0.81 for physical, self-evaluative, and social outcomes. Differences in outcome expectation scores between the intervention and control arms will be analyzed.
  This 5-point Likert scale contains 19 items with the outcome expectation score ranging from 19 to 95. A higher score indicates a higher expectation of doing physical activity for diverse health, cancer, social, and psychological outcomes.
Feasibility activity knowledge | Baseline, 3 months, 9 months
  Physical activity knowledge will be measured using a 5-point behavioral capacity Likert scale that assesses participants' knowledge about types, intensity, frequency, and skills of doing physical activity. The knowledge score ranges from 5 to 25. A higher score indicates a higher level of knowledge about doing appropriate physical activity. Differences in knowledge scores between the intervention and control arms will be analyzed.
Self-efficacy | Baseline, 3 months, 9 months
  Self-efficacy will be measured using a nine-item barrier self-efficacy scale and a four-item task self-efficacy scale to assess participants' confidence in overcoming barriers to physical activity and ability to do physical activity. The two self-efficacy scales have Cronbach's alpha of 0.96 and 0.89 among cancer patients, respectively. The total self-efficacy score ranges from The total self-efficacy score ranges from 13 to 65. A higher score indicates a higher level of confidence in overcoming barriers and doing physical activity. Differences in total self-efficacy scores between the intervention and control arms will be analyzed.
Physical activity engagement | Baseline, 3 months, 9 months
  Physical activity engagement is measured by a 6-point Likert scale that measures the habit strength for moderate-to-vigorous physical activity. The total habit score ranges from 17 to 102. A higher score indicates a greater engagement in physical activity. Differences in habit scores between the intervention and control arms will be analyzed.
Physical activity enjoyment | Baseline, 3 months, 9 months
  Enjoyment is measured by a short version of the Physical Activity Enjoyment Scale (4-item). The enjoyment score ranges from 4 to 20. A higher score indicates a higher level of enjoyment participants perceive from doing physical activity. Differences in enjoyment scores between the intervention and control arms will be analyzed.
Pain score | Baseline, 3 months, 9 months
  Pain will be measured using a 4-item 5-point Likert pain interference scale from the Patient-Reported Outcomes Measurement Information System (PROMIS) measures. The pain score ranges from 4 to 20. A higher score indicates a higher level of pain interfering with participants' activities. Differences in the pain score between intervention and control groups will be analyzed.
Fatigue score | Baseline, 3 months, 9 months
  Fatigue will be measured using a 4-item 5-point Likert fatigue scale from the PROMIS measures. The fatigue score ranges from 4 to 20. A higher score indicates a higher level of fatigue. Differences in the fatigue score between intervention and control groups will be analyzed.
Depression score | Baseline, 3 months, 9 months
  Depression will be measured using a 4-item 5-point Likert emotional distress scale from PROMIS measures. The depression score ranges from 4 to 20. A higher score indicates a higher level of depression. Differences in the depression score between intervention and control groups will be analyzed.
Bowel dysfunction score | Baseline, 3 months, 9 months
  Bowel dysfunction will be measured using a 5-point Likert scale from the PROMIS that measures gastrointestinal diarrhea and constipation. The bowel dysfunction score ranges from 15 to 75. A higher score indicates a higher gastrointestinal discomfort participants have. Differences in the score between intervention and control groups will be analyzed.
Sleep quality | Baseline, 3 months, 9 months
  Sleep quality will be measured using a 4-item 5-point Likert scale from the PROMIS measures. The sleep score ranges from 4 to 20. A higher score indicates a better sleep quality. Differences in the sleep score between intervention and control groups will be analyzed.
Neurotoxicity | Baseline, 3 months, 9 months
  Neurotoxicity will be measured using a 4-item 5-point Likert scale from the PROMIS measures. The neurotoxicity score ranges from 4 to 20. A higher score indicates greater neurotoxicity symptoms participants report. Differences in the neurotoxicity score between intervention and control groups will be analyzed.
Quality of life score | Baseline, 3 months, 9 months
  Quality of life score will be measured using the 36-item Short Form Health Survey. The quality of life score ranges from 0 to 100. The score for each item in the form ranges from 0 to 100 and the average scores of items representing general physical, mental, and social health are calculated, respectively. A higher score indicates better general physical, mental, or social health. Differences in the score between intervention and control groups will be analyzed.
Inflammation biomarkers level | Baseline, 3 months, 9 months
  Inflammation biomarkers, including IL-4, IL-10, IL-6, and TNF-α, will be measured by collecting participants' blood samples using the Dried Blood Spot card. The differences in inflammation biomarker levels between the intervention and control groups will be analyzed.
Dietary behaviors | Baseline, 3 months, 9 months
  Dietary behaviors are measured by the Rapid Eating Assessment for Participants (Shortened Version, 16 items). The diet score ranges from 1 to 46. A higher score indicates that the participant follows healthier dietary behaviors. Differences in diet scores between the intervention and control arms will be analyzed.
Comorbidities | Baseline, 3 months, 9 months
  Comorbidities will be measured using the Self-administered Comorbidity Questionnaire. Participants are asked to self-report whether they have or received treatment for 14 common health problems. The comorbidity score ranges from 0 to 28. Differences in comorbidity scores between the intervention and control arms will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Hirschey, Ph.D, RN, Principal Investigator — UNC Lineberger Comprehensive Cancer Center
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Hirschey R, Xu J, Woodard N, Duggins P, Lea DF, Milner JL, Coleman K Jr, Bryant AL, Sanoff HK, Triglianos T, Zou B, Burse NR, Hoover RL, Leeman J, Wheeler SB, Battaglini CL, Valle CG. Community-Engaged Approach to Increase Physical Activity Among Black Individuals With Colorectal Cancer: Protocol for a Feasibility Randomized Controlled Trial of the Physical Activity Centers Empowerment Study. JMIR Res Protoc. 2025 Oct 17;14:e65804. doi: 10.2196/65804. PMID 41105939
- See also: University of North Carolina Lineberger Comprehensive Cancer Center Clinical Trials — http://unclineberger.org/patientcare/clinical-trials/clinical-trials